CLINICAL TRIAL: NCT04241822
Title: Musculoskeletal Pain in Long-term Dizziness- Incidence, Prognosis and Measures
Brief Title: Musculoskeletal Pain in Long-term Dizziness
Acronym: MUPID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western Norway University of Applied Sciences (Other)
Collaborators: Haukeland University Hospital (Other)
Responsible Party: Principal Investigator, Liv Heide Magnussen, Professor, Western Norway University of Applied Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 6849
Record Dates: First submitted 2020-01-15; First posted 2020-01-27 (Actual); Last update posted 2024-08-07 (Actual); Status verified 2024-08

CONDITIONS: Vestibular Disease; Musculoskeletal Pain; Rehabilitation
Keywords: vestibular disease; musculoskeletal pain; prognosis; vestibular rehabilitation
MeSH Terms: conditions — Vestibular Diseases; Musculoskeletal Pain | interventions — Cognitive Behavioral Therapy; Exergaming

STUDY DESIGN:
Intervention Model Description: After 1 year participants who still have dizziness complaints will be offered one of two interventions:
  1. Group-based vestibular rehabilitation combining cognitive intervention, vestiular exercises and body awareness therapy
  2. Exergaming intervention with virtual reality exercises using data games and videos, and other balance exercises.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vestibular exercises combined with cognitive therapy (Experimental): The intervention is in groups of 8-10 patients. The interventions consists of cognitive therapy, vestibular exercises and body awareness therapy, 8 group sessions
  Interventions: Behavioral: Vestibular exercises combined with body awareness exercises and cognitive therapy
- Exergaming (Experimental): The intervention is individual and consist of non-immersive virtual reality exercises to improve balance
  Interventions: Behavioral: Exergaming

INTERVENTIONS:
Behavioral: Vestibular exercises combined with body awareness exercises and cognitive therapy — The intervention is group based and is a combination of information/education, vestibular exercises (head movements and gaze stability exercises) body awareness exercises and cognitive therapy
  Arms: Vestibular exercises combined with cognitive therapy
Behavioral: Exergaming — The intervention consists of different balance exercises using non-immersive virtual reality
  Arms: Exergaming

SUMMARY:
This project is aimed at patients with dizziness believed to be due to conditions in the balance organ in the inner ear (vestibular diseases). Dizziness can be bothersome and influence postural control negatively, and can cause secondary musculoskeletal disorders. Dizziness can also result in reduced work capacity. The purpose of the project is to strengthen the knowledge base regarding symptom burden, prognosis and treatment of prolonged dizziness. The hypothesis is that musculoskeletal pain at baseline is a prognostic factor for prolonged dizziness.

DETAILED DESCRIPTION:
Patients referred to an tertiary otorhinolarynglogical clinic due to dizziness will be invited to participate in the study. The aims are to examine the prevalence, extent and distribution of musculoskeletal pain in patients with prolonged dizziness, and to investigate the associations between musculoskeletal pain, dizziness symptoms, psychological and physical function and health-related quality of life.

Furthermore, the aim is to monitor the natural course of the dizziness symptoms and functional status in these patients, and examine risk factors for prolonged disability after 6 and 12 months. The hypothesis is that muscle pain and distress at baseline may be independently associated with prolonged complaints at follow-up.

Finally, patients who still are dizzy and have pain after 12 months will be invited to participate in one of two group interventions a) modified vestibular rehabilitation and b) virtual reality / exergaming. The interventions will be feasibility studies with a pre-post design.

ELIGIBILITY:
Inclusion Criteria:

* Patients referred to an otorhinolaryngological university clinic due to suspected vestibular disorders (dizziness)
* Patients must be bothered with dizziness at the time of consultation

Exclusion Criteria:

* Patients uable to fill in questionnaires due language barriers
* Patients not able to undergo diagnostic and testing procedures
* Patients with vestibular Schwannoma
* Patients with diving-related inner ear injuries

Ages: 18 Years to 67 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2020-08-15 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Dizziness Handicap Inventory. 0-100 (high score worst) | Baseline, 26 weeks, 1 year, through study completion, an average 18 months
  Baseline status and change in dizziness handicap

SECONDARY OUTCOMES:
Nordic Pain Questionnaire. 0-10 (high score worst) | Baseline, 26 weeks, 1 year, through study completion, an average 18 months
  Baseline status and change in musculoskeletal pain
Vertigo Symptom Scale. 0-60 (high score worst) | Baseline, 26 weeks, 1 year, through study completion, an average 18 months
  Baseline status and change in vertigo symptoms
RAND-12 health related quality of life. 0-60 (high score better) | Baseline, 26 weeks, 1 year
  Baseline status and change in health related quality of life
Hospital Anxiety and Depression Scale. 0-42 (high score worst) | Baseline, 26 weeks, 1 year
  Baseline status and change in anxiety and depression symptoms
Dizziness Catastrophising Scale. 0-52 (high score worst) | Baseline, 26 weeks, 1 year, through study completion, an average 18 months
  Baseline status and change in catastrophising thoughts about the dizziness
Posturography. Body sway while standing on a force platform. | Baseline,1 year, through study completion, an average 18 months
  Baseline status and change after intervention
Four tests of Body flexibility derived from the Global Physiotherapy Examination- 52 | Baseline,1 year, through study completion, an average 18 months
  Baseline status and change after intervention
Walking test preferred speed, 6 m (m/s) | Baseline,1 year, through study completion, an average 18 months
  Baseline status and change after intervention
Walking test fast speed, 6 m (m/s) | Baseline,1 year, through study completion, an average 18 months
  Baseline status and change after intervention
Grip Strength | Baseline
  Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Gro Anita F Flaten, ph.d., Study Director — Western Norway University of Applied Sciences; Evelyn Neppelberg, ph.d., Study Director — Haukeland University Hospital
Locations (1):
- Haukeland University Hospital, Bergen, Norway